CLINICAL TRIAL: NCT03312933
Title: Associated Joint Pain With CAM Walking Boot Wear
Brief Title: Associated Joint Pain With Controlled Ankle Movement (CAM) Walker Boot Wear
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jeremy Smith, Jeremy T Smith, MD., Principal Investigator, Instructor, Harvard Medical School, Brigham and Women's Hospital
Other Study IDs: 2015P000327/BWH
Record Dates: First submitted 2017-10-13; First posted 2017-10-18 (Actual); Results first posted 2019-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2018-08

CONDITIONS: Pain; Ankle Injuries
MeSH Terms: conditions — Pain; Ankle Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Duration of boot >2 weeks: All patients who were placed into a CAM walker boot for >2 weeks were prospectively enrolled. Patients were placed by an orthopedic cast technician into either a tall or short CAM walker boot, based upon the appropriate boot type needed for treatment. Inclusion criteria included anticipated boot wear for at least two weeks, and weightbearing as tolerated weightbearing restrictions. Exclusion criteria included transitioning into a CAM walker boot as part of a postoperative protocol, injury requiring restricted weightbearing, or an additional acute injury to the lower back or lower extremity. Those who subsequently reported wearing the boot for less than two weeks or had a treatment plan change were removed from the study.

SUMMARY:
This study evaluates the location, frequency and duration of secondary site pain relating to immobilization in a CAM walker boot.

DETAILED DESCRIPTION:
Patients wearing a CAM walker boot for treatment of a foot or ankle injury were prospectively enrolled and evaluated for new or worsened secondary site pain. Surveys at four time points were completed to evaluate the presence of secondary site pain, its severity, and its impact on overall function.

ELIGIBILITY:
Inclusion Criteria:

* All patients enrolled in the study must have an injury that requires wear of a CAM walking boot for at least two weeks and have ambulation ad libitum without other aids (e.g crutches, canes, scooters, wheelchairs, etc.).

Exclusion Criteria:

* Patients will be excluded from the study if they are a recent post-operative patient for lower extremity injury, have an additional acute injury to a lower extremity or back other than the foot or ankle injury being treated by the CAM walking boot at the time of initiation of treatment, have an ongoing or history of lower extremity joint injury, arthritis, or back pain or have restricted weightbearing as instructed by a physician (i.e. for ankle fracture that cannot weightbear).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who were placed into a CAM walker boot for >2 weeks were prospectively enrolled. Patients were placed by an orthopedic cast technician into either a tall or short CAM walker boot, based upon the appropriate boot type needed for treatment. Those who subsequently reported wearing the boot for less than two weeks or had a treatment plan change were removed from the study.
  Demographic information was gathered, including age, sex, race or ethnicity, body mass index (BMI), history of lower extremity or lower back injury, history of chronic pain (e.g. fibromyalgia, chronic opiate use, chronic regional pain syndrome), and cigarette smoking history. The diagnosis was recorded for which the CAM walker boot was required.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-03-19 (Actual); Primary Completion 2016-03-18 (Actual); Study Completion 2016-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy T Smith, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CAM Walker Boot for >2 Weeks: All patients who were placed into a CAM walker boot for >2 weeks were prospectively enrolled in the study. At the time of initiation of boot wear, patients were placed by an orthopedic cast technician into either a tall Aircast AirSelect Elite™ or short Aircast AirSelect™ CAM walker boot, based upon the diagnosis and appropriate boot type needed for treatment. Inclusion criteria included minimum age of 18 years, anticipated boot wear for at least two weeks, and weightbearing as tolerated weightbearing restrictions. Exclusion criteria included transitioning into a CAM walker boot as part of a postoperative protocol, injury requiring restricted weightbearing, or an additional acute injury to the lower back or lower extremity. Those who subsequently reported wearing the boot for less than two weeks were excluded. Additionally, patients who had a treatment plan change, such as proceeding with lower extremity surgery during the study period, were removed from the study.
Period: Overall Study
Arm/Group | CAM Walker Boot for >2 Weeks
Started | 100
Completed | 46
Not Completed | 54
Not completed — Protocol Violation | 15
Not completed — Lost to Follow-up | 36
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | CAM Walker Boot for >2 Weeks
Number analyzed (Participants) | 46
Age, Continuous [Mean (Full Range); unit: years] | 49 [22 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 39
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 46
Body Mass Index [Number; unit: participants] — A BMI was calculated for each patient. The were then separated into Normal (below 25 kg/m^2), Overweight (25-30 kg/m^2), and Obese (above 30 kg/m^2).
  participants
    Normal (below 25) | 24
    Overweight (25-30) | 10
    Obese (above 30) | 12
Injury Type [Count of Participants; unit: Participants]
  Fracture | 17
  Sprain | 7
  Tendon Problem | 17
  Other | 5
Secondary Site Pain [Count of Participants; unit: Participants]
  One or more secondary site pains | 27
  No secondary site pains | 19
Type of CAM walker boot [Count of Participants; unit: Participants]
  Tall CAM Boot | 31
  Short CAM Boot | 15

OUTCOME MEASURES:

1. Primary Outcome: The Presence and Severity of Secondary Site Pain
Description: The primary outcome was the presence of secondary site pain that developed or worsened during CAM walker boot wear. Surveys inquired about the presence of secondary site pain, defined as lower back, ipsilateral hip, contralateral hip, ipsilateral knee, contralateral knee, contralateral ankle, and contralateral foot. Severity of pain was assessed using a 100-point visual analog scale (VAS), with zero indicating no pain and 100 representing the worst pain imaginable.
Time Frame: At the time of transitioning out of the boot
Measure: Count of Participants; unit: Participants
Groups:
- Duration of CAM Walking Boot Wear >2 Weeks: All patients who were placed into a CAM walker boot for >2 weeks were prospectively enrolled in the study. At the time of initiation of boot wear, patients were placed by an orthopedic cast technician into either a tall Aircast AirSelect Elite™ or short Aircast AirSelect™ CAM walker boot, based upon the diagnosis and appropriate boot type needed for treatment. Inclusion criteria included minimum age of 18 years, anticipated boot wear for at least two weeks, and weightbearing as tolerated weightbearing restrictions. Exclusion criteria included transitioning into a CAM walker boot as part of a postoperative protocol, injury requiring restricted weightbearing, or an additional acute injury to the lower back or lower extremity. Those who subsequently reported wearing the boot for less than two weeks were excluded. Additionally, patients who had a treatment plan change, such as proceeding with lower extremity surgery during the study period, were removed from the study.
Arm/Group | Duration of CAM Walking Boot Wear >2 Weeks
Number analyzed (Participants) | 46
Participants | 31

ADVERSE EVENTS:
Time Frame: Patients were followed until three months after transitioning out of the boot.
Arm/Group | CAM Walker Boot for >2 Weeks
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes